CLINICAL TRIAL: NCT03431207
Title: Comparison of the Behavioral Dynamics Between Visually Impaired Infants and Healthy Controls
Brief Title: Behavioral Dynamics Between Infants With Visual Loss and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: CCPMOH2018-China-1
Record Dates: First submitted 2018-01-30; First posted 2018-02-13 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Behavioral Dynamics; Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- healthy group: For the "healthy" group, the visual acuity of both eyes was in the 95% referenced range with no structural abnormalities.
  The referenced range could be found in the following publication:
  Mayer, DL., et al. Monocular acuity norms for the Teller Acuity Cards between ages one month and four years. Investigative Ophthalmology & Visual Science. 36(3):671 (1995)
  Interventions: Other: Standardized video recording for behaviors
- mildly impaired group: The "mildly impaired" group was defined as a VA out of the 95% reference range in at least 1 eye, but the VA of both eyes was in the 99% referenced range with structural abnormalities.
  Interventions: Other: Standardized video recording for behaviors
- severely impaired group: For the "severely impaired" group, the VA of both eyes was out of the 99% referenced range or worse than light perception with structural abnormalities.
  Interventions: Other: Standardized video recording for behaviors

INTERVENTIONS:
Other: Standardized video recording for behaviors — A standardized apparatus, scenario, and procedure was applied to record all the behavioral phenotypes with minimized background interference and stimulation.
  For each standardized procedure, the guardian sits in the chair, holding the infant facing the stage. Each infant is given a few minutes to adapt to the surroundings and to be calm before recording. No hints or simulations are permitted during the entire process. The recording process lasted for over 5 minutes to ensure that behavioral phenotypes could be completely recorded.

SUMMARY:
An individual senses the world and reflects feedbacks via independent behaviors. Such precise collaboration of the sensory and behavioral systems is fundamental to survival and evolution. When a sensory modality is altered, the behavioral system has the potential to fit in a substitute modality. However, the specific dynamics of human behaviors in response to sensory loss remain largely unknown due to the paucities of representative situations and large-scale samples.

Here, the investigators focused on thousands of human infants who suffered varying degrees of visual stimuli deficiency in early stages, while their behavioral systems remained sensitive and thus retained high behavioral plasticity. Having access to this unique population provides an unprecedented opportunity to investigate the effect of diverse visual conditions on the behavioral system.

ELIGIBILITY:
Inclusion Criteria:

* Younger than 3 years of age

Exclusion Criteria:

* Any brain and mental illnesses, or other known illnesses that may affect the behavioral patterns

Max Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The investigators focused on thousands of human infants who suffered varying degrees of visual stimuli deficiency in early stages, while their behavioral systems remained sensitive and thus retained high behavioral plasticity. Having access to this unique population provides an unprecedented opportunity to investigate the effect of diverse visual conditions on the behavioral system.
Sampling Method: Non-Probability Sample
Enrollment: 4196 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Behavioral dynamics | baseline
  Eyeball movement (strabismus, nystagmus, and incongruous binocular movement); hand-related behaviors (eye rubbing, pressing, and poking); fixation-related behaviors (compulsive light gazing, compensatory head position, motionless fixation, and poor fixation); and eyelid reaction (frequent blinking, squint, and frown). Five experienced ophthalmologists identified the behaviors independently, and 2 professors with over 10 years of experience in pediatric ophthalmology department were consulted in cases of disagreement.

CONTACTS AND LOCATIONS:
Overall Officials: Yizhi Liu, Ph.D, Study Chair — Zhongshan Ophthalmic Center, Sun Yat-sen Univerisity
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Long E, Lin Z, Chen J, Liu Z, Cao Q, Lin H, Chen W, Liu Y. Monitoring and Morphologic Classification of Pediatric Cataract Using Slit-Lamp-Adapted Photography. Transl Vis Sci Technol. 2017 Nov 2;6(6):2. doi: 10.1167/tvst.6.6.2. eCollection 2017 Nov. PMID 29134133
- [Background] Japyassu HF, Malange J. Plasticity, stereotypy, intra-individual variability and personality: handle with care. Behav Processes. 2014 Nov;109 Pt A:40-7. doi: 10.1016/j.beproc.2014.09.016. Epub 2014 Sep 18. PMID 25241306